CLINICAL TRIAL: NCT03683628
Title: Treatment of Intermittent Claudication by G-CSF-mobilized Autologous Peripheral Blood Mononuclear Cells
Brief Title: Treatment of Intermittent Claudication by G-CSF-mobilized PB-MNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI016033012
Record Dates: First submitted 2018-09-03; First posted 2018-09-25 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Intermittent Claudication; PAD; Atherosclerotic Ischemic Disease
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor who measure the pain free walking distance, ABI, TBI,TCOM do not know the result of randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-MNC therapy (Active Comparator): The patientsin PB-MNC therapy group will be injected with G-CSF mobilized PB-MNC into calf or thigh muscle of ischemic limb, Aspirin 81 mg/day, cilostazol 200 mg/day and walking exercise 3 times per week.
  Interventions: Procedure: PB-MNC therapy
- No PB-MNC therapy (Active Comparator): In patients in No PB-MNC therapy, they will receive aspirin 81 mg/day, cilostazol 200 mg/day and walking exercise 3 times per week.
  Interventions: Drug: No PB-MNC therapy

INTERVENTIONS:
Procedure: PB-MNC therapy — The patients will receive subcutaneous injection of Granulocyte colony stimulating factor (G-CSF) for 3 day. The mononuclear cell will be collected by blood cell separator. The 120 cc of cell solution will be injected into calf or thigh of ischemic limb (1cc per site) with needle no. 25 gauge. Patients will receive ASA 81 mg once daily and walking exercise 3 times/ week
  Arms: PB-MNC therapy
Drug: No PB-MNC therapy — Patients will receive ASA 81 mg once daily and walking exercise 3 times/ week
  Arms: No PB-MNC therapy

SUMMARY:
This study will investigate the efficacy of G-CSF mobilized mononuclear cell injection of patients with PAD who presented with intermittent claudication. Forty PAD patients who presented with intermittent claudication will be randomized into 2 groups. The control group will be treated by medication and walking exercise 3 times/ week. The experiment group will be injected G-CSF mobilized mononuclear cell ,medication and walking exercise 3 times/ week. Ankle brachial index(ABI), Toe brachial index (TBI) and transcutaneous oxygen measurement will be evaluated at the day of randomization, 1 , 3, 6 and 12 months

DETAILED DESCRIPTION:
This study will investigate the efficacy of G-CSF mobilized mononuclear cell injection of patients with PAD who presented with intermittent claudication. Forty PAD patients who presented with intermittent claudication will be randomized into 2 groups. The control group will be treated by medication and walking exercise 3 times/ week. The experiment group will be injected G-CSF mobilized mononuclear cell ,medication and walking exercise 3 times/ week. Ankle brachial index(ABI), Toe brachial index (TBI) and transcutaneous oxygen measurement will be evaluated at the day of randomization, 1 , 3, 6 and 12 months in the control group and day of randomization, 1 , 3, 6 and 12 months after injection of PB-MNC in the experiment group. Pain free walking distance will be evaluated at the day of randomization, 1 , 3, 6 and 12 months by pedometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic arterial occlusive disease who presented with intermittent claudication

Exclusion Criteria:

* Recent myocardial infarction
* Severe valvular heart disease
* After organ transplantation
* Cardiomyopthy( EF< 25%)
* Liver failure
* Coagulopathy
* HIV
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain free walking distance | 3 month
  the maximum distance which patient could walk without pain

SECONDARY OUTCOMES:
Ankle brachial index (ABI) | 1,3,6,12 month
  Ankle brachial indexThe Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm. It has been shown to be a specific and sensitive metric for the diagnosis of Peripheral Arterial Disease (PAD)
Toe brachial index (TBI) | 1,3,6,12 month
  Toe brachial indexThe toe brachial index is the ratio between toe pressure and the highest of the two brachial pressures
Transcutaneous oxygen measurement (TCOM) | 1,3,6,12 month
  Transcutaneous oxygen measurement
36-Item Short Form Health Survey (SF36) | 1,3,6,12 month
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting.
Pain free walking distance | 1,6,12 month
  the maximum distance which patient could walk without pain

CONTACTS AND LOCATIONS:
Overall Officials: Nuttawut SERMSATHANASAWADI, MD, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No